CLINICAL TRIAL: NCT04564326
Title: Pericapsular Nerve Group Block Versus Fascia Iliaca Block for Pre- and Post-Operative Analgesia in Elderly Patients With Hip Fracture
Brief Title: PENG Block Versus Fascia Iliaca Block for Pre- and Post-Operative Analgesia in Elderly Patients With Hip Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Khaled Moustafa Magdy Nasr Mohamed, Principal Investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 6228/20-7-2020
Record Dates: First submitted 2020-09-20; First posted 2020-09-25 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Hip Fractures
Keywords: PENG block; Hip fracture; analgesia; Fascia Iliaca block; ultrasound; Fentanyl
MeSH Terms: conditions — Hip Fractures; Agnosia | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group C (Active Comparator): Patients will be assigned to receive opioids analgesia before spinal anesthesia in the form of intravenous fentanyl in a dose of 1mic/kg divided into two boluses with 5 minutes interval in between before positioning the patient for spinal anesthesia.
  Interventions: Drug: Fentanyl
- Group P (Experimental): Patients will be assigned to receive Pericapsular Nerve Group Block (PENG Block) before positioning the patient for spinal anesthesia.
  Interventions: Procedure: Pericapsular nerve Group block
- Group F (Experimental): Patients will be assigned to receive Fascia Iliaca Block (F.I Block) before positioning for spinal anesthesia.
  Interventions: Procedure: Facia Iliaca block

INTERVENTIONS:
Procedure: Pericapsular nerve Group block — Under ultrasound guidance a needle is inserted between the iliopectineal eminence and the iliopsoas muscle and tendon to block articular branches supplying the capsule of hip joint.
  Other Names: PENG block
  Arms: Group P
Procedure: Facia Iliaca block — Under ultrasound guidance a needle is inserted between the fascia iliaca and Psoas muscle to block the femoral, obturator and lateral cutaneous nerves.
  Other Names: FI block
  Arms: Group F
Drug: Fentanyl — Intravenous fentanyl in a dose of 1mic/kg divided into two boluses with 5 minutes interval in between.
  Other Names: Intravenous opioid
  Arms: Group C

SUMMARY:
Clinical controled trial to compare between pericapsular Nerve Group Block and Fascia Iliaca Block to find the best way to provide analgesia for elderly patients with hip fracture in the pre- and post-operative periods.

DETAILED DESCRIPTION:
Pain is a major problem that has to be dealt with in case of hip fracture, as it resembles an obstacle for examination, positioning for receiving neuroaxial anesthesia and postoperative mobility and physiotherapy.

With the introduction of ultrasound in regional anesthesia and peripheral nerve blocks, regional analgesia float to the surface as a substitute for opioids with less side effects. Of the many techniques to provide regional analgesia for hip fractures; fascia iliaca block was widely used with good results. In 2018 Pericapsular Nerve Group Block was introduced to provide regional analgesia for hip fractures with interesting results.

In this study the investigators are going to compare Pericapsular Nerve Group Block and Fascia Iliaca Block to find the best way to provide analgesia for elderly patients with hip fracture in the pre- and post-operative periods.

ELIGIBILITY:
Inclusion Criteria:

1. Patient acceptance.
2. Accepted mental state of the patient.
3. Gender: both sexes.
4. Age above 65 years old.
5. Body mass index 18.5-35 kg/m2.
6. ASA physical status II and III.
7. Unilateral hip fracture assigned for surgical fixation.
8. Expected duration of surgery ≤ 3 hours.

Exclusion Criteria:

1. Associated trauma or multiple fractures.
2. Peripheral neuropathy.
3. Coagulopathy.
4. Infection at site of injection.
5. Allergy to the drugs used in the study.
6. Advanced kidney, liver or heart disease.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Comparison between the analgesic effect of both Pericapsular Nerve Group block and Fascia Iliaca block with VAS score. | Baseline
  Analysis of Visual Analogue Pain Score for both PENG block and FI block before and after each block during rest and movement to compare between their analgesic effect. The Visual Analogue Pain score is done by drawing a 10cm vertical line on a piece of paper with its limits "no pain" (0) on one side and "extreme pain" (10) on the other side. The patient will be asked to point where the pain (he/she) experiences lies on the line.

CONTACTS AND LOCATIONS:
Overall Officials: Khaled M Mohamed, Master degree, Principal Investigator — Zagazig University

REFERENCES:
- [Background] Parker M, Johansen A. Hip fracture. BMJ. 2006 Jul 1;333(7557):27-30. doi: 10.1136/bmj.333.7557.27. No abstract available. PMID 16809710
- [Background] Kowark A, Rossaint R, Coburn M. General versus spinal anesthesia for the elderly hip fractured patient. Curr Opin Anaesthesiol. 2019 Feb;32(1):116-119. doi: 10.1097/ACO.0000000000000679. PMID 30543554
- [Background] Neuman MD, Silber JH, Elkassabany NM, Ludwig JM, Fleisher LA. Comparative effectiveness of regional versus general anesthesia for hip fracture surgery in adults. Anesthesiology. 2012 Jul;117(1):72-92. doi: 10.1097/ALN.0b013e3182545e7c. PMID 22713634
- [Background] Yun MJ, Kim YH, Han MK, Kim JH, Hwang JW, Do SH. Analgesia before a spinal block for femoral neck fracture: fascia iliaca compartment block. Acta Anaesthesiol Scand. 2009 Nov;53(10):1282-7. doi: 10.1111/j.1399-6576.2009.02052.x. Epub 2009 Jul 22. PMID 19650803
- [Background] Morrison SR, Magaziner J, McLaughlin MA, Orosz G, Silberzweig SB, Koval KJ, Siu AL. The impact of post-operative pain on outcomes following hip fracture. Pain. 2003 Jun;103(3):303-311. doi: 10.1016/S0304-3959(02)00458-X. PMID 12791436
- [Background] Morrison RS, Dickman E, Hwang U, Akhtar S, Ferguson T, Huang J, Jeng CL, Nelson BP, Rosenblatt MA, Silverstein JH, Strayer RJ, Torrillo TM, Todd KH. Regional Nerve Blocks Improve Pain and Functional Outcomes in Hip Fracture: A Randomized Controlled Trial. J Am Geriatr Soc. 2016 Dec;64(12):2433-2439. doi: 10.1111/jgs.14386. Epub 2016 Oct 27. PMID 27787895
- [Background] Helmerhorst GT, Vranceanu AM, Vrahas M, Smith M, Ring D. Risk factors for continued opioid use one to two months after surgery for musculoskeletal trauma. J Bone Joint Surg Am. 2014 Mar 19;96(6):495-9. doi: 10.2106/JBJS.L.01406. PMID 24647506
- [Background] Pasero C. Fentanyl for acute pain management. J Perianesth Nurs. 2005 Aug;20(4):279-84. doi: 10.1016/j.jopan.2005.03.007. No abstract available. PMID 16102709
- [Background] Scurrah A, Shiner CT, Stevens JA, Faux SG. Regional nerve blockade for early analgesic management of elderly patients with hip fracture - a narrative review. Anaesthesia. 2018 Jun;73(6):769-783. doi: 10.1111/anae.14178. Epub 2017 Dec 26. PMID 29278266
- [Background] Curatolo M. Regional anesthesia in pain management. Curr Opin Anaesthesiol. 2016 Oct;29(5):614-9. doi: 10.1097/ACO.0000000000000353. PMID 27137511
- [Background] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Background] Shin JJ, McCrum CL, Mauro CS, Vyas D. Pain Management After Hip Arthroscopy: Systematic Review of Randomized Controlled Trials and Cohort Studies. Am J Sports Med. 2018 Nov;46(13):3288-3298. doi: 10.1177/0363546517734518. Epub 2017 Oct 13. PMID 29028436
- [Background] Haines L, Dickman E, Ayvazyan S, Pearl M, Wu S, Rosenblum D, Likourezos A. Ultrasound-guided fascia iliaca compartment block for hip fractures in the emergency department. J Emerg Med. 2012 Oct;43(4):692-7. doi: 10.1016/j.jemermed.2012.01.050. Epub 2012 Apr 9. PMID 22494596
- [Background] Short AJ, Barnett JJG, Gofeld M, Baig E, Lam K, Agur AMR, Peng PWH. Anatomic Study of Innervation of the Anterior Hip Capsule: Implication for Image-Guided Intervention. Reg Anesth Pain Med. 2018 Feb;43(2):186-192. doi: 10.1097/AAP.0000000000000701. PMID 29140962
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Dolan J, Williams A, Murney E, Smith M, Kenny GN. Ultrasound guided fascia iliaca block: a comparison with the loss of resistance technique. Reg Anesth Pain Med. 2008 Nov-Dec;33(6):526-31. doi: 10.1016/j.rapm.2008.03.008. PMID 19258967
- [Background] Langley GB, Sheppeard H. The visual analogue scale: its use in pain measurement. Rheumatol Int. 1985;5(4):145-8. doi: 10.1007/BF00541514. PMID 4048757
- [Background] Wei LA, Fearing MA, Sternberg EJ, Inouye SK. The Confusion Assessment Method: a systematic review of current usage. J Am Geriatr Soc. 2008 May;56(5):823-30. doi: 10.1111/j.1532-5415.2008.01674.x. Epub 2008 Apr 1. PMID 18384586
- [Background] Ross VH, Pan PH, Owen MD, Seid MH, Harris L, Clyne B, Voltaire M, Eisenach JC. Neostigmine decreases bupivacaine use by patient-controlled epidural analgesia during labor: a randomized controlled study. Anesth Analg. 2009 Aug;109(2):524-31. doi: 10.1213/ane.0b013e31819518e4. Epub 2009 Apr 17. PMID 19377050
- See also: Quality-Based Procedures: Clinical Handbook for Hip Fracture. — http://www.hqontario.ca/evidence/publications-and-ohtac-recommendations/clinical-handbooks

DOCUMENTS (1):
  • Study Protocol (2020-08-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT04564326/Prot_000.pdf